CLINICAL TRIAL: NCT02736032
Title: Cryopreserved-thawed Embryo Transfer in Down or Non-down Regulated Hormonally Controlled Cycles: a Prospective, Randomized Study
Brief Title: Cryopreserved-thawed Embryo Transfer With or Without Gonadotropin Releasing Hormone Agonist
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Nile Ivf Center, Cairo, Egypt (Other); Kamal Shaeer center of infertility (Unknown)
Responsible Party: Principal Investigator, Yasmin Ahmed Bassiouny, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12016
Record Dates: First submitted 2016-03-30; First posted 2016-04-13 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer; Gonadotropin-Releasing Hormone; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With GnRHa (Active Comparator): Cryopreserved-thawed embryo transfer cycle, with endometrial preparation using GnRHa followed by external estradiol and progesterone. The GnRHa depot from will be given on day 21 of the preceding cycle, on day 1 of the transfer cycle, the patient will receive 6 mg/ day of estradiol followed up on day 12 of the cycle, if the endometrium is less than 8 mm, till day 15 of the cycle estradiol will be increased to 8 mg/day until 8 mm or more. Then, serum estradiol and progesterone levels are collected, and progesterone 800 mg vaginal suppository will be added and embryo transfer performed 2 to 3 days later.
  Interventions: Procedure: Embryo transfer; Procedure: Serum Estradiol and Progesterone levels; Drug: GnRH agonist; Drug: External Estradiol; Drug: Progesterone
- Without GnRHa (Active Comparator): Cryopreserved-thawed embryo transfer cycle, with endometrial preparation using external estradiol and progesterone only. On day 1 of the transfer cycle, the patient will receive 6 mg/ day of estradiol and followed up on day 12 of the cycle, if the endometrium did not reach 8 mm, till day 15 of the cycle the dose will be increased to 8 mg/day until the endometrium is 8 or more mm. When the endometrium is ready, serum estradiol and progesterone levels are collected, then progesterone 800 mg vaginal suppository will be added and embryo transfer performed 2 to 3 days later.
  Interventions: Procedure: Embryo transfer; Procedure: Serum Estradiol and Progesterone levels; Drug: External Estradiol; Drug: Progesterone

INTERVENTIONS:
Procedure: Embryo transfer — The transfer of cryopreserved-thawed embryos inside the uterus aiming to achieve pregnancy
Procedure: Serum Estradiol and Progesterone levels — Serum estradiol and serum progesterone levels in blood on the day of start of progesterone supplementation
Drug: GnRH agonist — GnRH agonist given on day 21 of the cycle preceding the embryo transfer
  Other Names: Decapeptyl SR
  Arms: With GnRHa
Drug: External Estradiol — Estradiol started on day1 of the cycle for endometrial prepartaion
  Other Names: estradiol valerate of Cycloprogenova tablets
Drug: Progesterone — progesterone as luteal phase support start after endometrium is well prepared
  Other Names: Cyclogest vaginal suppositories

SUMMARY:
Traditionally, the use of GnRH-a suppression was considered essential for adequate endometrial hormonal modulation in cryopreserved-thawed embryo transfer cycles. Several studies, however, have questioned its necessity for controlled endometrial preparation. Using a high dose of estradiol from day 1 of the cycle will suppress the gonadotroph, preventing folliculogenesis and excessive secretion of LH, allowing adequate endometrial preparation without GnRH-a.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 years
* BMI 20-30
* Regular menses.
* No PCOS, no endometriosis
* No uterine anomalies or lesions
* No severe male factor
* All grade 1 cleaved stage embryos

Exclusion Criteria:

* Less than 20 or more than 35 years
* BMI less than 20 or more than 30
* Irregular cycles
* PCOS or endometriosis
* Uterine anomalies or lesions
* Severe male factor
* Poor quality embryos for transfer
* Severe

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 5 weeks after embryo transfer]
  the detection of intrauterine gestational sac with positive pulsations
Live birth rate | 9 months
  Pregnancy ending with a live birth

SECONDARY OUTCOMES:
Estradiol and Progesterone levels on day of start of progesterone supplementation | 12 to 20 days
  The serum levels of estradiol and progesterone before embryo transfer
Endometrial thickness on day of start of progesterone supplementation | 12 to 20 days
  The endometrial thickness on the day of starting progesterone supplementation to transfer the embryos
Number of days needed for adequate (> 8mm) endometrial thickness | 12 to 20 days
  Number of days on external hormones to prepare endometrium
Cycle cancellation: not related to thawing, thin endometrium, high P. OR related to embryos not surviving thawing. | 12 to 20 days
  Cycle cancellation: not related to thawing, thin endometrium, high Progesterone. OR related to embryos not surviving thawing.
Chemical pregnancy rate | 14 days after embryo transfer
  positive serum Beta HCG 14 days after embryo transfer
Implantation rate. | 5 weeks after embryo transfer
  the ratio between the number of embryos transferred and the number of sacs
Early miscarriage rate | 3 months
  Pregnancy loss in the first 12 weeks gestation
Ongoing pregnancy rate | 3 months
  Pregnancy ongoing beyond 12 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Eman K Shaeer, MD, Study Director — Cairo University
Locations (3):
- Egypt (3):
  - IVF centre, Obstetrics and Gynaecology Department, Cairo University Hospitals (Kasr EL Aini), Cairo
  - Kamal Shaeer center of infertility, Giza
  - Nile IVF center, Giza

IPD SHARING:
Plan to Share IPD: Yes